CLINICAL TRIAL: NCT01568983
Title: The Effects of Polyphenol-rich Berry Juice on Blood Pressure and Additional CVD Related Parameters in Pre-hypertensive Subjects
Brief Title: The Effects of Polyphenol-rich Berry Juice on Blood Pressure in Hypertensive Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: Fellesjuice AS (Unknown); Nofima (Other)
Responsible Party: Principal Investigator, Rune Blomhoff, Professor, University of Oslo
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Optijuice
Record Dates: First submitted 2012-03-07; First posted 2012-04-02 (Estimated); Last update posted 2012-07-03 (Estimated); Status verified 2012-06

CONDITIONS: Pre-hypertension; Hypertension
MeSH Terms: conditions — Prehypertension; Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Placebo Comparator): 12 weeks intake of 0.5 liter/day placebo juice containing sugar, aromas and salt corresponding to the berry juices in the other groups.
  Blood pressure will be taken at time point 0,6 and 12 weeks. Blood and urine samples will be collected and weight and bioelectric impedance will be monitored at time point 0 and 12 weeks.
  Interventions: Dietary Supplement: Placebo
- Mana-juice (Active Comparator): 12 weeks intake of 0.5 liter/day of a commercially available berry juice (Mana blue) rich in polyphenols (grape, cherries, bilberries and aronia).
  Blood pressure will be taken at time point 0,6 and 12 weeks. Blood and urine samples will be collected and weight and bioelectric impedance will be monitored at time point 0 and 12 weeks.
  Interventions: Dietary Supplement: Mana-juice
- Optijuice (Active Comparator): 12 weeks intake of 0.5 liter/day of berry juice rich in polyphenols (grape, cherries, blueberry and aronia) and added extract from press cake of black currant.
  Blood pressure will be taken at time point 0,6 and 12 weeks. Blood and urine samples will be collected and weight and bioelectric impedance will be monitored at time point 0 and 12 weeks.
  Interventions: Dietary Supplement: Optijuice

INTERVENTIONS:
Dietary Supplement: Placebo — 500 ml/day Per 100g 6.25 g sucrose 6.25 g maltodextrin 1.3 g citric acid E330 (pH 3.0) 2.5 g Carmine solution E120 (4% carmine colouring agent) 0.025 g blueberry aroma Potassium sorbate E202 water
  Arms: Control
Dietary Supplement: Mana-juice — 500 ml/day of a grape,cherry, bilberry,aronia juice 13g carbohydrates/100g 150mg K/100g
  Arms: Mana-juice
Dietary Supplement: Optijuice — 500 ml/day of a Grape,cherry, bilberry,aronia, black current juice 13g carbohydrates/100g 150mg K/100g
  Arms: Optijuice

SUMMARY:
The purpose of this study is to investigate the effects of berry juices containing different levels of polyphenols on blood pressure and other cardiovascular risk factors.

The study is a 12 week double blinded randomized controlled intervention trial. The subjects will be divided in three groups where one receives a placebo juice while the two other will consume 0.5 liter of juice containing different levels of polyphenols. Blood pressure will be monitored and blood samples will be taken.

ELIGIBILITY:
Inclusion Criteria:

* Pre-hypertension or hypertension systolic blood pressure in the 130-179 mmHg range and/or diastolic blood pressure in the 85-109 mmHg range)
* BMI 20-35 kg/m2
* Stable weight (change <4 kg previous 12 weeks)

Exclusion Criteria:

* Regular use of blood pressure lowering agens
* Diabetes type I or II
* Smokers
* Allergy to grape, cherries, blueberries/bilberries, black currant, aronia
* Supplements for weight loss
* Changes in pharmacological treatment of hyperlipidemia or hyperglycemia (initiation, termination or changes in dosage) last 30 days prior to inclusion or during the study period (run-in and intervention)
* Participation in a drug trial during the previous 30 days

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2011-12; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Systolic and diastolic blood pressure | Screening, baseline, 6 and 12 weeks
  Change in blood pressure from baseline to 6 weeks and 12 weeks
Platelet aggregation | Baseline and 12 weeks
  Change in platelet aggregation from intervention start till end analyzed by PFA100.
Cardiovascular disease risk factors | Baseline and 12 weeks
  The effect of polyphenole-rich diet on cardiovascular disease risk factors in blood samples will be analyzed.
Diabetes related parameters in blood and urine | Baseline and 12 weeks
  The effect of different doses and types of polyphenoles on diabetes related biomarkers in blood and urine will be analyzed.
Blood cell expression of stress-response and CVD related genes | Baseline and 12 weeks
  Effect of polyphenole-rich diet on blood cell expression of stress-response and cardiovascular disease related genes by low density array and/or whole genome expression (microarray).

SECONDARY OUTCOMES:
Polymorphisms in cardiovascular disease related genes | Baseline
  Single nucleotide polymorphisms will be analyzed and eventually grouped and compared with the mentioned outcome measures to reveal individual mechanisms of the hypothetized effects of the intervention.
Whole genome transcription profiles and methylation patterns | Baseline and 12 weeks
  Effects of polyphenoles on transcription profiles and methylation pattern will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Rune Blomhoff, PhD, Principal Investigator — University of Oslo
Locations (1):
- University of Oslo, Oslo, Norway